CLINICAL TRIAL: NCT00109083
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging, Multicenter Study of the Efficacy of RWJ-333369 in the Prophylaxis of Migraine
Brief Title: A Study of the Efficacy of RWJ-333369 in the Prevention of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 333369-MIG-2001
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Migraine Headaches
Keywords: Migraine; Headaches; Migraine headaches; Head pain
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

INTERVENTIONS:
Drug: RWJ-333369

SUMMARY:
The purpose of this study is to evaluate whether RWJ-333369 is a safe and effective treatment in reducing the number of migraine headaches when added to a person's usual medications for acute migraine headache relief.

ELIGIBILITY:
Inclusion Criteria:

* Established history of migraines for at least 1 year;
* Have between 3 and 12 migraine attacks per month, and no more than 15 headache days in total per month;
* Migraines must have first started before age 50.

Exclusion Criteria:

* Most frequent headache type is not migraine;
* Failed 3 or more studies of effective migraine-preventing medications;
* Overuse of pain medications to treat migraines;
* Not willing to stop use of migraine-preventing medications;
* Significant serious concomitant diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the average monthly migraine frequency from the baseline period to the entire double-blind treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical R & D, L.L.C., Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (25):
- United States (25):
  - Northport, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Berkeley, California
  - Golden, Colorado
  - Miami, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Baton Rouge, Louisiana
  - Brockton, Massachusetts
  - Springfield, Massachusetts
  - Chaska, Minnesota
  - Springfield, Missouri
  - Greensboro, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Mogadore, Ohio
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - Richardson, Texas
  - Alexandria, Virginia
  - Olympia, Washington
  - Middleton, Wisconsin

REFERENCES:
- [Derived] Cady RK, Mathew N, Diener HC, Hu P, Haas M, Novak GP; Study Group. Evaluation of carisbamate for the treatment of migraine in a randomized, double-blind trial. Headache. 2009 Feb;49(2):216-26. doi: 10.1111/j.1526-4610.2008.01326.x. PMID 19222595